CLINICAL TRIAL: NCT06202144
Title: Physiological Effects of Personalized Noninvasive Support in Acute Hypoxemic Respiratory Failure
Brief Title: Personalized Noninvasive Support in Acute Hypoxemic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5173-2
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Acute Hypoxic Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Noninvasive support (Experimental): Helmet noninvasive support, with positive end-expiratory pressure (PEEP)=12 cmH2O and the minimal pressure-support level capable of generating inspiratory effort between 5 and 10 cmH2O
  Interventions: Device: Noninvasive support
- Continuous positive airway pressure (Active Comparator): Helmet CPAP will be delivered through a high-flow generator and PEEP valve set at 12 cmH2O
  Interventions: Device: Noninvasive support
- Noninvasive ventilation (Active Comparator): Helmet NIV will be delivered in the pressure-support mode, with PEEP=12 cmH2O and pressure support=12 cmH2O
  Interventions: Device: Noninvasive support

INTERVENTIONS:
Device: Noninvasive support — Noninvasive respiratory support delivered through a helmet

SUMMARY:
The optimal noninvasive respiratory support for acute hypoxemic respiratory failure is debated. Recent preliminary data indicate that both pressure-support noninvasive ventilation (NIV) and continuous-positive airway pressure (CPAP) may be of benefit. While often applied interchangeably in clinical practice, NIV and CPAP have different effects on the inspiratory effort, which is the major determinant of self-inflicted lung injury. Also, inspiratory effort widely varies among individuals.

The purpose of this study is to assess the physiological effects of a noninvasive respiratory support approach guided by inspiratory effort, as compared to CPAP and NIV, in patients with moderate-to-severe acute hypoxemic respiratory failure.

DETAILED DESCRIPTION:
Patients with acute hypoxemic respiratory failure will undergo a decremental pressure-support trial during helmet noninvasive support. The following pressure-support settings will be applied sequentially, with positive end-expiratory pressure kept constant and equal to 10-12 cmH2O: 20 cmH2O, 16 cmH2O, 12 cmH2O, 8 cmH2O and high-flow-driven CPAP. Inspiratory effort will be monitored during the trial through esophageal manometry. The personalized setting of noninvasive support will be defined as the minimal pressure-support level capable of generating inspiratory effort between 5 and 10 cmH2O.

Personalized noninvasive support will be then compared to conventionally-set NIV and CPAP in a randomized cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypoxemic respiratory failure and PaO2/FiO2<200 mmHg
* PaCO2<45 mmHg
* Respiratory failure not caused by exacerbation of chronic pulmonary disease, cardiac failure or fluid overload

Exclusion Criteria:

* Pregnancy
* Contraindication to helmet support
* Contraindication to esophageal manometry
* Contraindication to electrical-impedance tomography monitoring
* Recent surgery involving the abdomen or the thorax
* Pneumothorax or documented barotrauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Tidal volume | 1 hour
  Tidal volume size, assessed with electrical impedance tomography
Transpulmonary driving pressure | 1 hour
  The positive inspiratory swing in transpulmonary pressure, calculated as airway pressure minus esophageal pressure

SECONDARY OUTCOMES:
Inspiratory effort | 1 hour
  Inspiratory effort, defined as the negative deflection in esophageal pressure
Respiratory rate | 1 hour
  Respiratory rate per minute
Blood oxygenation | 1 hour
  PaO2/FiO2 ratio
Work of breathing | 1 hour
  Simplified esophageal pressure pressure-time product
Corrected minute ventilation | 1 hour
  Minute ventilation (assessed with electrical impedance tomography) normalized to PaCO2
Tidal volume distribution | 1 hour
  Tidal volume distribution in the four lung regions of interest (ventral, mid-ventral, mid-dorsal and dorsal), assessed with electrical impedance tomography
End-expiratory lung impedance | 1 hour
  End-expiratory lung impedance, assessed with electrical impedance tomography
Pendelluft extent | 1 hour
  Pendelluft, assessed with electrical impedance tomography and expressed in % of tidal volume size
Lung compliance | 1 hour
  Defined as the ration of tidal volume to transpulmonary driving pressure
Dyspnea | 1 hour
  Dyspnea, defined through a visual analog scale ((ranging from 0 to 10, with representing most severe dyspnea)

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Luca Grieco, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon reasonable request